CLINICAL TRIAL: NCT01802047
Title: Milk Volume Production in Mothers of Preterm Infants: Electric Pumping Modalities
Brief Title: Impact of Different Electric Pumping Modalities on Milk Volume Production in Mothers of Preterm Infants
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: d/t changes in routine modality of milk expression by electric pump.
Sponsor: Tel-Aviv Sourasky Medical Center (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Supportive Care
Other Study IDs: TASMC-13-SD-0678-12-CTIL
Record Dates: First submitted 2013-02-19; First posted 2013-03-01 (Estimated); Last update posted 2016-03-29 (Estimated); Status verified 2016-03

CONDITIONS: Prematurity
Keywords: Mothers of Preterms; Breastfeeding Mothers of Preterm infants; mother milk feeding
MeSH Terms: conditions — Premature Birth

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Electric Pump Modality (Experimental): Each mother follows all 3 electric pump modalities in a randomized order.
  Interventions: Procedure: milk expression with electric pump

INTERVENTIONS:
Procedure: milk expression with electric pump
  Other Names: Medella Electric breast pump

SUMMARY:
Initiating and sustaining breastfeeding are common challenges in neonatal units.

It is known that hindmilk expressed at the end of the expression session has a higher fat content.

Previous studies have shown that simultaneous pumping is more effective at producing milk than sequential pumping. However this approach is often felt uncomfortable by the mothers, and sequential pumping is preferred.

The purpose of this study is to determine which modality of milk expression by electric pump is the most efficient and productive when sequential pumping is used.This is done by assessing the milk volume expressed per expression and its macronutrients content.

DETAILED DESCRIPTION:
The study will last for 6 days. Each mother will express breast milk following two designed modalities in a random fashion, for two days each.

The two designed modalities are:

1. Complete pumping of one breast (first left) for 15 min, followed by complete pumping of the right breast for 15 min, until the breast is empty.
2. Pumping both breast simultaneously for 15 min.

At day one of the study, the mothers will follow the standard pumping modality in practice at our department.

In between the two studied procedures at day 4 of the study, the mothers will again follow the standard pumping modality.

On each day of the study, in the morning after the first expression of the day, a sample of 2 ml of pumped breastmilk will be taken, and the total volume of the daily expressed milk will be recorded.

ELIGIBILITY:
Inclusion Criteria:

* Mothers of Preterms

Exclusion Criteria:

* HIV infected mothers

Ages: 18 Years to 60 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 0 (Actual)
Dates: Start 2013-08; Primary Completion 2017-12 (Estimated); Study Completion 2018-12 (Estimated)

PRIMARY OUTCOMES:
Daily volume of expressed breast milk under a specific electric pumping modality | after 15 minutes of electric expression of each breast
  The total volume of all milk expression sessions of the day will be recorded. This, for each 6 days of the study.

SECONDARY OUTCOMES:
Composition of expressed milk under a specific electric pumping modality | after the first morning session of electric milk expression
  Fat, Protein and Carbohydrate concentrations will be assessed after each morning session of milk expression by using the mid-infrared milk analyzer (Miris AB, Uppsala, Sweden)

CONTACTS AND LOCATIONS:
Overall Officials: Shaul Dollberg, MD, Principal Investigator — Tel Aviv Medical Center
Locations (1):
- Department of Neonatology Tel Aviv Medical Center, Tel Aviv, Israel